# Deciphering Patient Participation: Insights from Observational Data in Scleroderma Clinical Trials

An Informed Consent Form For Power Clinical Trial's

Observational Study Involving Patients in Scleroderma Clinical

Trials

Date: February 9, 2024

### Introduction

Have you considered participating in a clinical trial for scleroderma? Understanding why individuals choose to join, stay involved, or opt out of these trials is crucial for maximizing their impact.

This invitation introduces you to our observational study seeking to answer this very question. Your participation, entirely voluntary and withdrawable at any time, holds significant value.

What does participating entail? Primarily completing questionnaires and participating in brief follow-up calls, designed to minimize any potential risks. While direct personal benefits may not be immediate, your contribution will fuel groundbreaking research to optimize clinical trial experiences for the scleroderma community.

By uncovering the key factors influencing participation, we aim to develop more effective recruitment strategies and enhance patient engagement, ultimately leading to better treatment options and outcomes for individuals like you.

Before making your decision, we encourage you to thoroughly review the consent form and discuss any concerns with our research team, healthcare providers, or any trusted confidants. Remember, your informed choice is paramount.

## **Understanding Your Choices in Clinical Trials**

Clinical trials play a pivotal role in unlocking new treatment options for scleroderma, but questions remain regarding the inclusivity of participants. This research delves into the factors that influence your decisions about joining, leaving, or rejoining scleroderma clinical trials. Understanding these motivators is crucial for creating research experiences that are more relevant and enriching for everyone.

We are committed to recruiting a diverse group of participants to ensure our findings accurately reflect the experiences of a wider population. We aim to uncover how factors like age, race, income level, and education shape your decisions about participating in clinical trials. This knowledge will be used to develop more effective strategies to engage individuals from historically underrepresented groups in future trials.

Your participation in this study is entirely voluntary, and you have the right to withdraw at any point without facing any consequences. The study involves minimal risk and primarily entails completing questionnaires and participating in follow-up phone calls. We encourage you to carefully review the consent form and ask any questions you may have.

By participating in this study, you will play a critical role in shaping the future of scleroderma research. By understanding your choices, we can work together to develop more inclusive and effective research experiences that ultimately lead to better treatments for this challenging condition.

# Risks and Safeguards in Scleroderma Observational Studies

Observational studies of scleroderma offer valuable insights without involving experimental treatments. However, it's essential to understand potential risks before making an informed decision about participation. These may include data privacy concerns, emotional distress stemming from the study topic, and rare but possible adverse events from study procedures.

To ensure you fully understand the potential risks and benefits, carefully review the informed consent document and engage in open dialogue with the research team. They are committed to providing comprehensive information and addressing any questions or concerns you may have.

The research team prioritizes participant safety and has implemented robust safeguards to minimize risks. Data privacy is of paramount importance, and measures are in place to protect your information. Additionally, support is available to address any emotional distress that may arise.

Remember, participation is entirely voluntary, and you can withdraw at any time without penalty. Should you experience any concerns or discomfort, the research team is readily available to provide assistance and ensure your well-being.

## **Exploring Factors Affecting Your Participation in Clinical Trials**

Clinical trials offer valuable opportunities for medical progress, but it's essential to understand the possibility of early termination. Sponsors or researchers may halt the trial due to various reasons, such as lack of funding, concerns about participant safety, or revised understanding of the research question.

Similarly, your participation might end due to personal circumstances like unexpected health changes, pregnancy, emerging information prompting you to reconsider, or difficulty following study procedures. Open communication and careful consideration of these possibilities before enrolment are crucial.

Transparency is paramount throughout the research process. The informed consent document outlines potential reasons for early termination, alongside the expected timeline and your rights as a participant. If you have any questions or concerns, the research team is available to discuss them thoroughly.

Remember that even if unexpected circumstances lead to early termination, your voice matters. You retain the right to withdraw at any time, with or without reason, and without penalty. The research team remains committed to open communication and addressing any questions or concerns you may have throughout the trial.

## This Study Compared to Other Scleroderma Clinical Trials

Participation in scleroderma clinical studies is solely at your discretion, and you retain the right to withdraw at any point without facing repercussions.

Take an active role in exploring available <u>scleroderma research</u> options by utilizing Clinicaltrials.gov, a comprehensive database managed by the National Institutes of

Health (NIH). This resource grants you access to information on numerous active studies worldwide, offering the ability to refine your search based on your unique location and medical needs.

Furthermore, Power's reference page provides a regularly updated list of ongoing scleroderma clinical trials actively seeking participants. Leverage these tools to actively engage in the research process and make informed choices about your possible involvement.

Remember, you are at the center of this decision. Carefully consider the available information, pose any questions you may have to healthcare professionals, and ultimately choose the path that best aligns with your personal goals and preferences.

#### Online Resources on Inclusive Clinical Trials

Unveiling the complexities and opportunities surrounding diversity in clinical trials is crucial for advancing medical research. Thankfully, a wealth of online resources offers valuable insights. Here are two noteworthy articles:

El-Galaly, Tarec Christoffer, Verena I. Gaidzik, Mihnea-Alexandru Gaman, Darko Antic, Jessica Okosun, Mhairi Copland, Veronika Sexl et al. "A Lack of Diversity, Equity, and Inclusion in Clinical Research Has Direct Impact on Patient Care." *HemaSphere* 7, no. 3 (2023).

Hurd, Thelma C., Charles D. Kaplan, Elise D. Cook, Janice A. Chilton, Jay S. Lytton, Ernest T. Hawk, and Lovell A. Jones. "Building trust and diversity in patient-centered oncology clinical trials: an integrated model." *Clinical Trials* 14, no. 2 (2017): 170-179.

By engaging with these resources, researchers, healthcare professionals, and patients alike can gain valuable knowledge and work together to ensure that clinical trials truly represent the diverse communities they aim to serve.

# Participant Acknowledgement

By providing your signature on this consent form, you become an active participant in the research process, acknowledging and agreeing to the following:

- You have taken the time to carefully read and fully comprehend this informed consent document. We encourage you to engage in open dialogue with us and explore alternative viewpoints to ensure your decision is well-informed.
- All your inquiries regarding the research project and its methods have been satisfactorily addressed, leaving you confident and equipped to participate.
- You have thoroughly considered the potential benefits, drawbacks, and alternative options associated with your involvement in the research.
- Your voluntary participation in this study will not jeopardize your legal rights in any way.
- We are committed to maintaining open communication and promptly informing you of any significant updates that could affect your decision to continue participating in the research.
- Signing this consent form allows you to raise any remaining questions or concerns you may have before proceeding.

By acknowledging these key commitments, we embark on this research journey together, fostering an environment of shared responsibility and mutual respect.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| Name of Participant | Signature of Participant | Date |

#### Researcher's Declaration

As the researcher, I recognize my role in facilitating the patient's informed decision-making. Through thorough explanations and open dialogue, I have ensured the patient possesses a comprehensive understanding of the study and its implications. Additionally, we have explicitly confirmed the voluntary nature of their participation, placing their autonomy at the center of this research partnership.

By working together to ensure informed consent, we empower the patient to participate actively and confidently in the research journey.

| Signature of Researcher Who Re | eceived Consent | |
|--------------------------------|---------------------------|------|
| Name of Investigator | Signature of Investigator | Date |